CLINICAL TRIAL: NCT02986698
Title: A Single-Center, Non-Randomized Study of the Safety and Efficacy of in Utero Hematopoietic Stem Cell Transplantation for the Treatment of Fetuses with Alpha Thalassemia Major
Brief Title: In Utero Hematopoietic Stem Cell Transplantation for Alpha-thalassemia Major (ATM)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment ended early due to interim data suggesting a lack of efficacy. Interim data did demonstrate that IUHSCT was safe and well tolerated, but the PI and DSMB agreed that enrollment should not continue under the current treatment protocol.
Sponsor: University of California, San Francisco (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Tippi Mackenzie, Professor of Surgery, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-21157
Record Dates: First submitted 2016-12-05; First posted 2016-12-08 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Alpha Thalassemia Major; Hemoglobinopathy; with Thalassemia; Hemoglobinopathies; Fetal Anemia; Fetal Hydrops; Alpha; Thalassemia; Thalassemia Major; Thalassemia Alpha; A-Thalassemia
Keywords: intrauterine transfusion; in utero human stem cell transplantation
MeSH Terms: conditions — Thalassemia; Hemoglobinopathies; Hydrops Fetalis; alpha-Thalassemia; beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- in utero hematopoietic stem cell transplantation (Experimental): Perform in utero hematopoietic stem cell transplantation at the time of intrauterine transplantation in fetuses with alpha-thalassemia major. The cellular product is: Semi-allogeneic, Related, Maternal Bone Marrow-Derived, Miltenyi CliniMACS Plus enriched CD34+ hematopoietic stem cells administered in utero at a dose of 1 x 10^7-10^9 cells/kg fetal weight with equal to or less than 1% CD3+ T cells (equivalent to 10^5-10^7 T cells/kg fetal weight) in a final volume of 2-5ml suspended in 5% human serum albumin in Normosol buffer (Hospira, Inc.).
  Stem cells will be administered immediately before the red blood cells intravenously via the umbilical vein during the clinically indicated IUT. All participants will receive one dose of stem cells but may receive additional transfusions as clinically indicated.
  Interventions: Biological: in utero hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: in utero hematopoietic stem cell transplantation — This is a phase 1 safety study to demonstrate it is safe for both the mother and fetus to perform In utero hematopoietic stem cell transplantation of maternal derived stem cells at the time of intrauterine transplantation of red blood cells to treat fetuses affected with alpha-thalassemia major.

SUMMARY:
The investigators aims to evaluate the safety of in utero hematopoietic stem cell transplantation in fetuses with alpha-thalassemia major performed at the time of in utero transfusion of red blood cells.

DETAILED DESCRIPTION:
Alpha thalassemia major (ATM) is almost universally fatal in utero and represents an orphan disease with an unmet need for effective therapies. The only current treatment to allow the fetus to be born is to perform in utero transfusions (IUT) of red blood cells to treat the anemia and avoid the complications of hydrops and fetal demise. Often, affected pregnancies undergo elective termination after diagnosis. Cases with prenatal diagnosis of ATM who receive IUT and survive to birth will ultimately require lifelong monthly blood transfusions or bone marrow transplant, if a suitable donor is identified.

This is a phase 1 clinical trial to demonstrate the safety, feasibility and efficacy of performing in utero stem cell transplantation on fetuses affected with ATM. The investigators aim to recruit ten participants with a prenatal diagnosis of ATM. Participants will undergo bone marrow harvest and an in utero transfusion combined with maternal stem cells. Transplanting maternal cells into the fetus takes advantage of existing maternal-fetal tolerance during pregnancy. Hematopoietic stem cell (HSC) transplantation into the fetus takes advantage of the developing fetal immune system to induce tolerance to the transplanted cells without using conditioning or immunosuppression. Performing stem cell transplantation at the same time as IUT minimizes any additional procedural risk to the fetus.

The investigators hope to demonstrate that it is safe and feasible to perform in utero stem cell transplantation. Additionally, the investigators want to demonstrate postnatal chimerism of maternal cells so that, if a bone marrow transplant remains necessary after delivery, conditioning and immune suppression will not be required.

ELIGIBILITY:
Inclusion Criteria:

* Male or female fetuses from 18 weeks and 0/7 days to 26 weeks 0/7 days gestation with a diagnosis of alpha-thalassemia major by chorionic villus sampling (CVS), amniocentesis, cordocentesis or by identification of parents as genetic carriers, and identification of fetal anemia or signs of impending hydrops, for whom parents elect to pursue in utero transfusion, and are willing to undergo subsequent IUT for the remainder of gestation.
* parents must consent to fetal autopsy in the event of a fetal demise
* adequate bone marrow harvest from maternal participant is a condition for inclusion

Exclusion Criteria:

* Fetal Subject Exclusion Criteria: Fetal participants will be excluded if they have a second major anatomic anomaly (not related to the underlying thalassemia) that contributes a significant morbidity or mortality risk, or echocardiogram or ultrasound findings that indicate a high risk of fetal demise after fetal intervention.
* Maternal Subject Exclusion Criteria: Maternal participants will be excluded if they have one or more morbidities that would preclude bone marrow harvest and fetal intervention including, but not limited to, morbid obesity with BMI > 35, maternal cardiac disease, mirror syndrome, symptomatic maternal anemia, or if they develop preterm premature rupture of membranes (PPROM) or active preterm labor (PTL).

Ages: 18 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Maternal participant tolerance of bone marrow harvest | 5 year recruitment phase to include time of bone marrow harvest through 30 days after delivery
  Maternal participant tolerance of bone marrow harvest defined as not requiring interventions for preterm labor, bleeding, infection or prolonged hospitalization.
Safety of in utero hematopoietic stem cell transplantation when performed at the same time as in utero blood transfusion for the fetal participant | 5 year recruitment plus 1 year data collection phase to include time of IUHCT through 1 year after delivery
  safety for fetal participant defined by survival 24 hours after procedure, fetal survival till birth, neonatal survival through discharge of hospitalization and no evidence of graft versus host disease

SECONDARY OUTCOMES:
Adequate bone marrow harvest from the maternal participant | 5 year recruitment phase
  This is defined as approximately 200-300 cc of bone marrow from which 10^7-10^9 CD34+ cells/kg fetal weight with 10^5-10^7 CD3+ cells/kg fetal weight will be isolated.
successful engraftment | 5 year recruitment plus data collection phase to include time of IUHCT through 1 year after delivery
  The primary efficacy endpoint is successful engraftment of maternal bone marrow- derived CD34+ hematopoietic stem cells measured by establishment of maternal participant donor cell chimerism equal to or greater than 1% donor cells in the circulation of the fetal recipient. Chimerism will be determined in cord blood at birth, or at a corrected gestational age of 40 weeks, if there is preterm delivery, followed weekly for the first 4 weeks of life, and monthly for one year in the infant to monitor the stability of engraftment.

CONTACTS AND LOCATIONS:
Overall Officials: Tippi Mackenzie, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreger EM, Singer ST, Witt RG, Sweeters N, Lianoglou B, Lal A, Mackenzie TC, Vichinsky E. Favorable outcomes after in utero transfusion in fetuses with alpha thalassemia major: a case series and review of the literature. Prenat Diagn. 2016 Dec;36(13):1242-1249. doi: 10.1002/pd.4966. Epub 2016 Dec 7. PMID 27862048
- [Background] Derderian SC, Jeanty C, Walters MC, Vichinsky E, MacKenzie TC. In utero hematopoietic cell transplantation for hemoglobinopathies. Front Pharmacol. 2015 Jan 12;5:278. doi: 10.3389/fphar.2014.00278. eCollection 2014. PMID 25628564
- [Background] Vichinsky E. Advances in the treatment of alpha-thalassemia. Blood Rev. 2012 Apr;26 Suppl 1:S31-4. doi: 10.1016/S0268-960X(12)70010-3. PMID 22631041
- [Background] MacKenzie TC. Fetal Surgical conditions and the unraveling of maternal-fetal tolerance. J Pediatr Surg. 2016 Feb;51(2):197-9. doi: 10.1016/j.jpedsurg.2015.10.059. Epub 2015 Nov 4. PMID 26653947
- [Background] MacKenzie TC, David AL, Flake AW, Almeida-Porada G. Consensus statement from the first international conference for in utero stem cell transplantation and gene therapy. Front Pharmacol. 2015 Feb 10;6:15. doi: 10.3389/fphar.2015.00015. eCollection 2015. No abstract available. PMID 25713535
- [Background] Jeanty C, Derderian SC, Mackenzie TC. Maternal-fetal cellular trafficking: clinical implications and consequences. Curr Opin Pediatr. 2014 Jun;26(3):377-82. doi: 10.1097/MOP.0000000000000087. PMID 24759226
- [Background] Nijagal A, MacKenzie TC. Clinical implications of maternal-fetal cellular trafficking. Semin Pediatr Surg. 2013 Feb;22(1):62-5. doi: 10.1053/j.sempedsurg.2012.10.011. PMID 23395148
- [Background] Nijagal A, Flake AW, MacKenzie TC. In utero hematopoietic cell transplantation for the treatment of congenital anomalies. Clin Perinatol. 2012 Jun;39(2):301-10. doi: 10.1016/j.clp.2012.04.004. Epub 2012 May 8. PMID 22682381
- [Background] Nijagal A, Wegorzewska M, Le T, Tang Q, Mackenzie TC. The maternal immune response inhibits the success of in utero hematopoietic cell transplantation. Chimerism. 2011 Apr;2(2):55-7. doi: 10.4161/chim.2.2.16287. PMID 21912720
- [Derived] Borges B, Canepa E, Chang IJ, Herzeg A, Lianoglou B, Kishnani PS, Harmatz P, MacKenzie TC, Cohen JL. Prenatal Delivery of Enzyme Replacement Therapy to Fetuses Affected by Early-Onset Lysosomal Storage Diseases. Am J Med Genet C Semin Med Genet. 2025 Sep;199(3):203-217. doi: 10.1002/ajmg.c.32132. Epub 2025 Jan 31. PMID 39891377